CLINICAL TRIAL: NCT03878940
Title: A Feasibility Study of Direct Access to a Newly Developed Abdominal ´Yes-No´ Pathway for Primary Care Patients With Vague and Non-specific Abdominal Symptoms
Brief Title: A Feasibility Study of Direct Access to an Abdominal ´Yes-No´ Pathway for Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16/2019
Record Dates: First submitted 2019-02-27; First posted 2019-03-18 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Cancer; Primary Health Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary care patients (Other): All GPs in the municipality of Silkeborg will be invited to participate. Any patient can be referred to the abdominal ´yes-no´ pathway, independently of their willingness to give one´s consent.
  Interventions: Diagnostic Test: Abdominal ´yes-no´ pathway

INTERVENTIONS:
Diagnostic Test: Abdominal ´yes-no´ pathway — A set of blood samples, a FIT, and an abdominal US (and a TVUS in women)

SUMMARY:
Background To optimise cancer outcome in Denmark, cancer diagnostic pathways should, beside cancer patient pathways (CPP) for alarm symptoms, also include a pathway for patients with vague and non-specific symptoms. Research has demonstrated that 50% of all cancers do not qualify for specific CPPs, although the majority of patients initially present symptoms in general practice.

Hypothesis Direct access to an abdominal 'yes-no' pathway is feasible in general practice. Aim The aim of this study is to assess the implementation and clinical implications of direct access to an abdominal 'yes-no' pathway for primary care patients with vague and non-specific abdominal symptoms Materials and methods The study is a feasibility study in which all general practitioners (GPs) in the municipality of Silkeborg in Central Denmark Region are offered direct access to a newly developed abdominal ´yes-no´ pathway for both men and women aged 30 years or above, who present vague and non-specific abdominal symptoms in primary care. The abdominal ´yes-no´ pathway consists of: 1) Medical and objective examination, 2) Selected blood samples and a Fecal Immunochemical test (FIT), and 3) Abdominal ultrasound (US) and transvaginal US (TVUS) (for women).

Perspectives This study will provide important knowledge on how to improve abdominal cancer diagnostics in general practice.

DETAILED DESCRIPTION:
Background Danish cancer patients have poorer cancer outcome compared to other European cancer patients. Earlier cancer diagnosis is a pivotal step to improve the prognosis, and there seems to be opportunity for improvement, as e.g. colon cancer is more often diagnosed at an advanced stage in Denmark than in other countries.

In Denmark, more than 11,500 abdominal cancers are registered yearly, which corresponds to 31% of all newly diagnosed cancers. The majority (75-85%) of cancer patients initially present symptoms to their GP. But only half of the patients present an alarm symptom, while 20% present serious non-specific symptoms, and 30% present vague non-specific symptoms. Site-specific CPPs for alarm symptoms were implemented in Denmark in 2008/2009 to optimise the diagnostic route for cancer. In 2012, a new Danish CPP was implemented to target patients with serious non-specific symptoms and signs of cancer (NSSC-CPP). No pathway exists for patients with vague abdominal symptoms.

Presenting in general practice with abdominal symptoms is very common. Most abdominal symptoms presented in general practice can be signs of serious disease in the abdomen and the pelvic region. However, in most cases, the symptoms are benign, self-limiting and harmless. Still, more than ten different cancer types can cause these symptoms, but clinically it is often difficult to distinguish between the symptoms.

For patients presenting vague symptoms to the GP, the ideal strategy could be easy and direct access to relevant investigations rather than a wait-and-see approach or referral to a CPP.

Aim The study sets out to investigate the need for an abdominal 'yes-no' pathway for primary care patients with vague and non-specific abdominal symptoms, how it could be clinically organised and integrated, and whether such pathway is feasible.

Material and methods Prior to the current intervention, a developmental part was conducted in 2018. It consisted of focus group meetings with 16 selected specialist, with expertise regarding patients with abdominal symptoms in general practice and abdominal cancers and other abdominal diseases.

The investigators assembled two focus groups during autumn 2017, each comprising the following experts: two GPs, a physician with expertise in gastroenterology, an abdominal surgeon, a radiologist, a gynecologist, a microbiologist and a physician in clinical biochemistry. The focus groups aimed to develop and agree on an abdominal 'yes-no' pathway using the following criteria: 1) reduce the time to diagnosis, 2) avoid unnecessary tests, 3) increase patient safety and minimise missed opportunities, 4) order the specific investigations temporally, 5) place responsibility and develop a structure and 6) illustrate an optimal pathway.

From January to September 2018, the investigators completed two meetings in each focus group, after which the investigators compared the results and gathered the groups in a common session. From the literature and the preliminary results of an yet unpublished register study, the investigators were able to present the clinical challenges to the participants during the meetings. Moreover, the possible access to investigations was presented (laboratory tests, imaging, endoscopies and access to specialist advice). Based on discussions during the meetings, the investigators developed an abdominal ´yes-no´ pathway. The abdominal ´yes-no´ pathway consists of three steps; 1) Medical and objective examination, 2) Selected blood samples and a FIT, and 3) Abdominal US and TVUS. The GP continues to hold responsibility for follow-up, while hospital examinations are performed on an outpatient basis with direct access from general practice. After finished investigation, the results from the tests will all return electronically to the referring GP.

The intervention is planned to initiate as a feasibility study at Silkeborg Regional Hospital from 1 April 2019. Agreements have been made with the hospital management, and an information meeting has taken place in March 2019 at the hospital. All GPs in the municipality of Silkeborg were invited to participate. An illustration, to hand out for involved GPs has been developed. Prior to investigation, all patients referred to the abdominal ´yes-no´ pathway will receive a consent form with information of the study. The inclusion period is 6 months from 1 April 2019 to 30 September 2019, after which the investigators will monitor the patients for up to 6 months.

The study has been approved and is registered in the Record of Processing Activities at the Research Unit of General Practice in Aarhus in accordance with the provisions of the General Data Protection Regulation (GDPR). The Central Denmark Region Committees on Health Research Ethics has concluded that the study can be conducted without an approval from the Committees (Request 16/2019). Further, The committee on multi-practice studies under the Danish College of General Practitioners (DSAM) and the Organisation of General Practitioners in Denmark (PLO) have been asked to recommend GPs to participate in the study.

The analyses will be descriptive with frequencies and incidence rates of use of the pathway corrected for practice population. An overview of all findings in the abdominal 'yes-no' pathway will be provided, and possible side effects will be assessed.

Perspectives The study will provide new important knowledge of patients with vague and non-specific abdominal symptoms, who do not fulfil access criteria for the CPPs, but for whom the diagnosis of an abdominal cancer should not be missed. This may improve the diagnostics of abdominal cancers or other serious abdominal disease in the future, aiming to reduce time to diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* GPs in the municipality of Silkeborg can refer patients with the following criteria to Silkeborg Regional Hospital:

Men and women ≥30 years old presenting with vague and non-specific abdominal symptoms for at least 3-4 weeks

Exclusion Criteria:

* Men or women who fulfil access criteria for the CPPs.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
The proportion of general practices using the abdominal 'yes-no' pathway | 6 months
  In the municipality of Silkeborg, 23 general practices will be offered direct access to the abdominal 'yes-no' pathway.
Number of patients referred to the abdominal 'yes-no' pathway | 6 months
  The number of patients referred to the abdominal 'yes-no' pathway, both overall from all 23 general practices in the municipality of Silkeborg, and per general practice. We expect one eligible patient from each GP every third week.
Indications used for requesting the abdominal 'yes-no' pathway | 6 months
Health care use within 6 months of intervention | 6 months
  'Health care use´ is defined as consultations, imaging and endoscopies performed in both primary and secondary care. Data will be collected through the Danish National Patient Registry and the Danish National Health Service Register.

SECONDARY OUTCOMES:
Number of patients with a diagnosis of cancer or another serious disease in the abdomen | 6 months
  Data from The Danish Pathology Register will be used to investigate for cancer diagnoses and other serious diseases up to 6 months after the diagnostics performed through the abdominal ´yes-no´ pathway.
Number of patients with unintended side effects | 6 months
  Number of patients with unintended side effect in consequence of the diagnostics performed in and caused by the abdominal 'yes-no' pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vedsted, Study Director — Research Unit of General Practice, Aarhus, Denmark; Henry Jensen, Study Chair — Research Unit of General Practice, Aarhus, Denmark; Henning Gronbaek, Study Chair — Dept. of Hepatology and Gastroenterology, Aarhus University Hospital, Denmark; Henning Glerup, Study Chair — Diagnostic Center, Silkeborg Regional Hospital, Denmark; Nanna Holt Jessen, Principal Investigator — Research Unit of General Practice, Aarhus, Denmark
Locations (1):
- Silkeborg Regional Hospital, Central Denmark Region, Silkeborg, Denmark